CLINICAL TRIAL: NCT02465671
Title: Prognostic Value of Plasma Thrombospondin-1 Levels After Acute Intracerebral Hemorrhage：A Pilot Study
Brief Title: Prognostic Value of Plasma Thrombospondin-1 Levels After Acute Intracerebral Hemorrhage
Status: Completed | Type: Observational
Sponsor: Jinhua People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Jhh2015024
Record Dates: First submitted 2015-06-04; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Cerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All blood samples from the patients at admission were collected in the separator tubes and centrifuged within 30 minutes at 1,000*g for 15 minutes. The plasma was removed and frozen at -70°C until measurement.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients group: All patients with acute spontaneous basal ganglia hemorrhage admitted to the Jinhua People's Hospital within the first 24 h from stroke during the same period were enrolled.

SUMMARY:
The current study was designed to investigate the change of plasma thrombospondin-1 levels and assess the prognostic predictive effect of plasma thrombospondin-1 levels in the patients with acute intracerebral hemorrhage.

DETAILED DESCRIPTION:
Thrombospondin-1 acts as an anti-angiogenic factor and its expression in rat brain is upregulated after intracerebral hemorrhage. The current study was designed to investigate the change of plasma thrombospondin-1 levels and assess the prognostic predictive effect of plasma thrombospondin-1 levels in the patients with acute intracerebral hemorrhage. About 110 patients will be recruited. All blood samples from the patients at admission were collected. Thrombospondin-1 levels in plasma were measured using sandwich immunoassays. The patients will be followed up till 6 months after intracerebral hemorrhage. The relationships between plasma thrombospondin-1 levels and 1-week mortality, 6-month mortality, 6-month overall survival, 6-month unfavorable outcome (modified Rankin Scale score >2) and disease severity reflected by hematoma volume and National Institutes of Health Stroke Scale score were assessed using multivariate analysis. It is proposed that elevated plasma thrombospondin-1 levels are independently associated with disease severity and clinical outcomes. It will be suggested thrombospondin has potential to be a good prognostic biomarker of intracerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* acute spontaneous basal ganglia hemorrhage admitted to the Jinhua People's Hospital within the first 24 h from stroke.

Exclusion Criteria:

* previous ischemic or hemorrhagic stroke, severe head trauma, use of antiplatelet or anticoagulant medication, presence of other prior systemic diseases including autoimmune diseases, uremia, liver cirrhosis, malignancy, and chronic heart or lung disease, recent infection (within a month), a surgical procedure and missing of follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with acute spontaneous basal ganglia hemorrhage admitted to the Jinhua People's Hospital within the first 24 h from stroke were enrolled.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
mortality after intracerebral hemorrhage | Follow-up of 6 months

SECONDARY OUTCOMES:
Unfavorable outcome (modified Rankin Scale score >2 ) | Follow-up of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Yu CHENG, Study Chair — Jinhua People's Hospital